CLINICAL TRIAL: NCT04782531
Title: Variations of Portal Flow During the Respiratory Cycle in Healthy Volunteers
Acronym: RESPIFLUX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2020_843_0150
Record Dates: First submitted 2021-03-02; First posted 2021-03-04 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Amplitude; Portal Blood Flow; MRI; Echo Planar Imaging
Keywords: Respiratory amplitude; Portal Blood Flow; MRI; Echo Planar Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: peripheral ECG — Subjects will be placed in supine position. The systematic use of a headset will reduce the noise inherent to the machine. A cardiac synchronization system using peripheral ECG allows the synchronization with the subject's heart rate.
Other: Standard MRI — Standard MRI examination using a torso coil consists of morphological and phase-contrast flow sequences(standard and EPI acquisitions).

SUMMARY:
The analysis of portal vein blood flow is important when assessing the severity and progression of liver disease. It is important to understand normal liver regulation in order to appreciate the evaluation of the effect of treatment during the disease progression. The influence of respiration on hepatic hemodynamics is still poorly understood, although some studies have shown a significant impact. The purpose of this project is to quantify the blood flow variations in the portal vein at different positions during the respiratory cycle by using a fast MRI sequence and an Echo Planar (EPI) acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans
* Healthy subject without history of hepatic disease

Exclusion Criteria:

* history of hepatic pathology
* pregnant woman
* claustrophobia
* major obesity
* any contraindication to MRI exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
flow rates variation between the fast sequence averaged values and the standard sequence | 30 minutes
  flow rates variation between the fast sequence averaged values and the standard sequence during free breathing.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No